CLINICAL TRIAL: NCT06265792
Title: A Randomized Controlled Trial to Explore the Efficacy of Stellate Ganglion Block in Obstructive Sleep Apnea
Brief Title: Efficacy of Stellate Ganglion Block in Obstructive Sleep Apnea
Acronym: OSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0125
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy.The experimental group was given Stellate Ganglion Block.
  Interventions: Behavioral: routine rehabilitation treatment; Procedure: Stellate ganglion block
- The control group (Active Comparator): All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy.
  Interventions: Behavioral: routine rehabilitation treatment

INTERVENTIONS:
Behavioral: routine rehabilitation treatment — All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy
Procedure: Stellate ganglion block — The patients were provided with Stellate ganglion block , using 0.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: The experimental group

SUMMARY:
The goal of this clinical trial is to test the efficacy of stellate ganglion block in Obstructive Sleep Apnea. The main question it aims to answer are:

• Can stellate ganglion block improve Obstructive Sleep Apnea? Patients were randomly divided into two groups, all provided with routine therapy. Based on this, the experimental group was given stellate ganglion block. The video fluoroscopic swallowing study was done to test the swallowing function before and after the study.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea is of increasingly high prevalence.

The goal of this clinical trial is to test the efficacy of stellate ganglion block in Obstructive Sleep Apnea. The main question it aims to answer are:

• Can stellate ganglion block improve Obstructive Sleep Apnea? Patients were randomly divided into two groups, all provided with routine therapy. Based on this, the experimental group was given stellate ganglion block. The video fluoroscopic swallowing study was done to test the swallowing function before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years diagnosed with OSA by polysomnography
* Patients with moderate to severe OSA (AHI > 15 events per hour)
* Patients who have undergone continuous positive airway pressure (CPAP) treatment for at least 3 months but have not achieved satisfactory therapeutic effects
* Patients who voluntarily agree to receive stellate ganglion block (SGB) treatment and sign the informed consent form

Exclusion Criteria:

* Patients with a history of allergy or contraindications to local anesthetics or corticosteroids
* Patients with severe cardiovascular, cerebrovascular, respiratory, hepatic, or renal diseases
* Patients with a history of neck surgery or cervical spine disease
* Patients with psychiatric disorders or other medical conditions that may affect the safety or effectiveness of SGB treatment
* Pregnant or lactating women
* Patients who have participated in other clinical trials within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale | day 1 and day 20
  This scale measures daytime sleepiness. By scoring the level of sleepiness in different situations, it can help evaluate whether a patient has OSA or other sleep disorders.Scores range from 0-24. Higher scores indicate more severe daytime sleepiness.

SECONDARY OUTCOMES:
Apnea-Hypopnea Index | day 1 and day 20
  Apnea-Hypopnea Index is a method to evaluate the severity of OSA. It calculates the number of apnea and hypopnea events per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Doctor, Study Chair — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Center Rehabilitation Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No